CLINICAL TRIAL: NCT06179251
Title: KNOW HOW TO POSITION THE SACCULE AND UTRICULE IN SCANNING: INTEREST IN INTRAVESTIBULAR DISLOCATIONS OF PISTONS OR CALIPER
Brief Title: KNOW HOW TO POSITION THE SACCULE AND UTRICULE IN SCANNING
Acronym: Luxation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8488
Record Dates: First submitted 2023-12-11; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Otosclerosis
Keywords: Otosclerosis; Vestibular dysfunction; Membranous Labyrinth
MeSH Terms: conditions — Otosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Titanium pistons cause MRI artifacts that prevent interpretation of the vestibule. This disadvantage is not present on CT but the vestibule is not visible. Hence the interest in creating a model with 6 reference cuts in order to position the utricle and the saccule in the vestibule in CT. Furthermore, the scanner has fewer contraindications, greater availability and a shorter examination time than MRI.

DETAILED DESCRIPTION:
The aim of the study is to analyze six normal sections chosen as reference in histology, high resolution T2 MRI and CT in order to compare them with precise topographical landmarks to position the posterior membranous labyrinth in CT. Then, apply the investigators' observations to cases of operated otosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old) and minors (≥ 6 years old)
* Subject having received an MRI of the internal ear canals from the HUS between 01/01/2018 and 01/01/2021 or a CT scan of the rocks between 07/01/2015 and 01/01/2021
* Normal MRI or CT on the side opposite the pathology.
* Normal tonal audiogram on the side opposite the pathology (peripheral facial paralysis assumed to be cold for MRI and petrous fracture for CT).
* Subject who has not expressed his opposition, after information, to the reuse of his data for the purposes of this research.
* Holders of authority who have not expressed their opposition, after information, to the reuse of their child's data for the purposes of this research

Exclusion Criteria:

* Subject having expressed opposition to participating in the study
* Holders of parental authority who have expressed their opposition to the reuse of their child's data for the purposes of this research
* Imaging with artifacts
* Absence of pure-tone audiogram or its abnormality on the side of the ear studied
* Any malformation or pathology of the vestibule on imaging on the side of the ear studied
* Subjects under guardianship or curatorship

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults (≥18 years old) and minors (≥ 6 years old) having received an MRI of the internal ear canals from the HUS between 01/01/2018 and 01/01/2021 or a CT scan of the rocks between 07/01/2015 and 01/01/2021
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of the anatomical structure referenced in the investigators' reading grid on each of the 6 predefined MRI or CT sections | up to 10 month

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Radiologie - CHU de Strasbourg - France, Strasbourg, France